CLINICAL TRIAL: NCT02567591
Title: Adapted Physical Activity Effect on Aerobic Function and in Patients in Pre Liver Transplantation
Acronym: FAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I15017 FAPA
Record Dates: First submitted 2015-09-29; First posted 2015-10-05 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2018-09

CONDITIONS: Motor Activity
Keywords: pre liver transplantation patients
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: physical activity program (Experimental): at home physical activity program (during 12 weeks)
  Interventions: Other: Physical activity
- B: conventional management (No Intervention): conventional management

INTERVENTIONS:
Other: Physical activity — walk (three times per week) and muscle building twice per week with the use of elastic bands. They will include 5 strengthening exercises mobilizing large muscle groups of the lower limbs (abs (if possible for the patient), hamstrings, quadriceps, triceps sural and gluteus maximus).
  Arms: A: physical activity program

SUMMARY:
Physical exercise has been identified as a major beneficial factor in the management of patients suffering from many chronic diseases especially cancer and in the context of cardiac or pulmonary transplantation. It contributes to an improvement of the quality of life and decreases treatment side effects and mortality. Aerobic fitness is constantly altered in cirrhotic patients and correlated to the severity of the hepatic disease. Moreover, in this setting, other etiological factors may be added like chronic obstructive bronchitis and alcoholic cardiomyopathy. In this population, muscle abnormalities with fatigue and cramps have been described. Muscle weakness in this condition may be comparable to that described in patients with chronic obstructive bronchitis and contributes to the decrease of aerobic fitness. Different causes such as muscle deconditioning, hypoxemia, denutrition, anti-rejection drugs increase this phenomenon after liver transplantation. Finally, the aerobic capacity or VO2max is a prognostic factor for survival and is linked to the number and the length of hospitalizations after liver transplantation (LT).

Therefore, physical activity is a valid and relevant way to improve quality of life, increase survival, and limit costs of hospitalizations. The aim of this study is to assess the effects of a personalized physical activity retraining program on aerobic capacity, strength and fatigue, in a population awaiting liver transplantation.

Purpose: The hypothesis is that an at home adapted retraining program conducted before LT, and including physical activity (aerobic and strength training), will improve aerobic fitness, peripheral strength, quality of life and decrease the hospitalization length in intensive care unit after LT.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 70 years of age,
* Signed informed consent,
* Medical indication to LT whatever the cause of the liver disease

Exclusion Criteria:

* Inability to understand the instructions of the trial,
* Patients who are subject to a court protection, wardship or guardianship order,
* Uncontrolled cardiac disease and ventricular ejection fraction (vef) < 50 %,
* Any other serious conditions which are not stabilized and in which physical exercise is contra-indicated,
* Pregnancy or suckling,
* Patients transplanted in extreme emergency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-11 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
VO2 max at 12 weeks | at 12 weeks
  To evaluate the impact of a personalized physical activity program after 12 weeks of exercise on the aerobic capacity measured by VO2 max, in patients awaiting liver transplantation.

SECONDARY OUTCOMES:
6 minutes walk test at week 12 | at 12 weeks
  To evaluate at Week 12: 6 minutes walk test
After liver transplantation: aerobic capacity (VO2 max) | 3 and 6 months after liver transplantation
  To evaluate after liver transplantation: aerobic capacity (VO2 max) 3 and 6 months after LT

CONTACTS AND LOCATIONS:
Overall Officials: Marilyne DEBETTE-GRATIEN, Principal Investigator — University Hospital, Limoges
Locations (2):
- France (2):
  - Limoges Hospital, Limoges
  - Tours hospital, Tours